CLINICAL TRIAL: NCT04779879
Title: A Multicenter, Randomized, Double-Blind, Parallel Group Phase II Study to Evaluate the Safety, Tolerability and Pharmacokinetics of a Second Generation VIR-7831 Material in Non-Hospitalized Participants With Mild to Moderate Coronavirus Disease 2019 (COVID-19)
Brief Title: Safety, Tolerability and Pharmacokinetics of Second Generation VIR-7831 Material in Non-hospitalized Participants With Mild to Moderate COVID-19
Acronym: COMET-PEAK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIR-7831-5006; GSK Study 216912 (Other: GlaxoSmithKline)
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Covid19
Keywords: SARS-CoV-2; coronavirus; coronavirus disease 2019; COVID-19
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — sotrovimab; DNA-(Apurinic or Apyrimidinic Site) Lyase

STUDY DESIGN:
Masking Description: Part A is double-blinded. Parts B and C are open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sotrovimab (Gen1) (Active Comparator): Part A (double-blinded) participants will be randomized to receive 500 mg of an IV infusion of Sotrovimab Gen 1 material or 500 mg of an IV infusion of VIR-7831 Gen 2 material
  Interventions: Biological: Sotrovimab (Gen1); Biological: Sotrovimab (Gen2)
- Sotrovimab (Gen2) (Active Comparator): Part B (open-label) participants will be randomized to receive 500 mg of Sotrovimab Gen2 material by IV infusion or by IM injection
  Part C (open-label) participants will be randomized to receive 500 mg of Sotrovimab Gen2 material by IV infusion or 250 mg by IM injection
  Interventions: Biological: Sotrovimab (Gen2)

INTERVENTIONS:
Biological: Sotrovimab (Gen1) — Participants will be randomized to receive an IV infusion of Sotrovimab Gen 1 material
  Arms: Sotrovimab (Gen1)
Biological: Sotrovimab (Gen2) — Participants will be randomized to receive Sotrovimab Gen2 material by IV infusion or by IM injection
  Arms: Sotrovimab (Gen2)
Biological: Sotrovimab (Gen2) — Participants will be randomized to receive Sotrovimab Gen2 material by IV infusion
  Arms: Sotrovimab (Gen1)

SUMMARY:
This is a phase 2 study in which subjects with coronavirus disease 2019 (COVID-19) will receive VIR-7831 (Sotrovimab) Generation 1 (Gen1) or VIR-7831 (Sotrovimab) Generation 2 (Gen2) and will be assessed for safety, tolerability, and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* For Part A, participants must be aged 18 years or older at the time of obtaining informed consent
* For Parts B and C, participants must be aged between 18 years and 69 years old at the time of obtaining informed consent
* Participants who have a positive SARS-CoV-2 test result ≤7 days prior to enrollment and oxygen saturation ≥94% on room air and have COVID-19 symptoms and ≤7 days from onset of symptoms

Exclusion Criteria:

* Currently hospitalized or judged by the investigator as likely to require hospitalization in the next 24 hours
* Symptoms consistent with severe COVID-19
* Participants who, in the judgement of the investigator are likely to die in the next 7 days.
* Severely immunocompromised participants
* For Parts A and B, prior receipt of a SARS-CoV-2 vaccine at any time prior to enrollment (vaccination with an authorized or approved SARS-CoV-2 vaccine will not be allowed for 90 days after dosing)
* For Parts B and C, conditions that would prohibit receipt of IM injections in the investigator's opinion
* For Parts A, B and C, receipt of any vaccine within 48 hours prior to enrollment (vaccination with an authorized or approved SARS-CoV-2 vaccine will not be allowed for 90 days after dosing)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (15):
  - Investigative Site, Anniston, Alabama
  - Investigative Site, Bakersfield, California
  - Investigative Site, Northridge, California
  - Investigative Site, Ft. Pierce, Florida
  - Investigative Site, Gainesville, Florida
  - Investigative Site, Hialeah, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, Orlando, Florida
  - Investigative Site, Pembroke Pines, Florida
  - Investigative Site, Tampa, Florida
  - Investigative Site, Columbus, Georgia
  - Investigative Site, Winfield, Illinois
  - Investigative Site, Rockville, Maryland
  - Investigative Site, The Bronx, New York
  - Investigative Site, Houston, Texas
- Canada (2):
  - Investigative Site, Sarnia, Ontario
  - Investigative Site, Toronto, Ontario
- Investigative Site, Milan, Italy
- Investigative Site, Daejeon, South Korea
- Spain (8):
  - Investigative Site, Alicante
  - Investigative Site, Barcelona
  - Investigative Site, Centelles
  - Investigative Site, Granada
  - Investigative Site, La Roca del Vallès
  - Investigative Site, Madrid
  - Investigative Site, Pozuelo de Alarcón
  - Investigative Site, Vigo

REFERENCES:
- [Derived] Gupta A, Perez-Rodriguez MT, Gonzalez-Rojas Y, Ramgopal M, Free A, Han J, Moore J, Givens N, Yates PJ, Walker JT, Connolly MB, Schnell G, Imber V, Anselm R, Winograd L, Segal S, Harrison S, Skingsley A, Aldinger M, Peppercorn A, Moya J. Safety, Tolerability, Pharmacokinetics, and Viral Pharmacodynamics of the Monoclonal Antibody Sotrovimab Administered via Intramuscular Injection in Participants with Early, Mild-to-Moderate COVID-19: A Randomized Clinical Trial. Drugs R D. 2025 Dec;25(4):353-365. doi: 10.1007/s40268-025-00529-2. Epub 2025 Nov 24. PMID 41284195
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized, parallel group study conducted in non-hospitalized participants with mild to moderate Coronavirus Disease 2019 (COVID-19) who received Sotrovimab (VIR-7831) Generation1 (Gen 1) and Gen2.
Pre-assignment Details: Total of 354 participants (30 participants in Part A, 167 participants in Part B, 157 participants in Part C) were enrolled in the study.
Groups:
- Part A-Sotrovimab Gen1: 500 mg IV: Participants received Sotrovimab (VIR-7831) Gen1 500 milligrams (mg) intravenous (IV) infusion on Day 1 in Part A.
- Part A- Sotrovimab Gen2: 500 mg IV: Participants received Sotrovimab (VIR-7831) Gen2 500 mg IV infusion on Day 1 in Part A.
- Part B- Sotrovimab Gen2: 500 mg IV: Participants received Sotrovimab (VIR-7831) Gen2 500 mg IV infusion on Day 1 in Part B.
- Part B- Sotrovimab Gen2: 500 mg IM: Participants received Sotrovimab (VIR-7831) Gen2 500 mg intramuscular (IM) injection on Day 1 in Part B.
- Part C- Sotrovimab Gen2: 500 mg IV: Participants received Sotrovimab (VIR-7831) Gen2 500 mg IV infusion on Day 1 in Part C.
- Part C- Sotrovimab Gen2: 250 mg IM: Participants received Sotrovimab (VIR-7831) Gen2 250 mg IM injection on Day 1 in Part C.
Period: Part A: Up to Week 24
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Started | 8 | 22 | 0 | 0 | 0 | 0
Treatment Received | 8 | 22 | 0 | 0 | 0 | 0
Completed | 8 | 22 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B: Up to Week 36
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Started | 0 | 0 | 84 | 83 | 0 | 0
Treatment Received | 0 | 0 | 84 | 82 | 0 | 0
Completed | 0 | 0 | 84 | 81 | 0 | 0
Not Completed | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Randomized, but did not receive treatment | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Period: Part C: Up to Week 36
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Started | 0 | 0 | 0 | 0 | 79 | 78
Treatment Received | 0 | 0 | 0 | 0 | 79 | 78
Completed | 0 | 0 | 0 | 0 | 75 | 75
Not Completed | 0 | 0 | 0 | 0 | 4 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM | Total
Number analyzed (Participants) | 8 | 22 | 84 | 82 | 79 | 78 | 353
Age, Customized [Count of Participants; unit: Participants] — Safety Population consisted of all randomized participants who were exposed to study intervention.
  Participants
    Participants: <=18 years | 0 | 1 | 0 | 1 | 0 | 0 | 2
    Participants: 19-64 years | 8 | 20 | 80 | 76 | 77 | 74 | 335
    Participants: >=65 years | 0 | 1 | 4 | 5 | 2 | 4 | 16
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population consisted of all randomized participants who were exposed to study intervention.
  Participants
    Female | 5 | 10 | 45 | 42 | 39 | 42 | 183
    Male | 3 | 12 | 39 | 40 | 40 | 36 | 170
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Safety Population consisted of all randomized participants who were exposed to study intervention.
  Participants
    Participants: Black or African American | 2 | 1 | 4 | 1 | 7 | 9 | 24
    Participants: White - White/Caucasian/European Heritage | 6 | 21 | 62 | 64 | 66 | 63 | 282
    Participants: White - Arabic/North African Heritage | 0 | 0 | 5 | 0 | 6 | 5 | 16
    Participants: Asian - East Asian Heritage | 0 | 0 | 2 | 2 | 0 | 0 | 4
    Participants: Asian - South East Asian Heritage | 0 | 0 | 11 | 13 | 0 | 0 | 24
    Participants: Asian - Central/South Asian Heritage | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Participants: American Indian Or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Participants: Mixed Asian Race | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With All Adverse Events (AEs) and Serious Adverse Events (SAEs) Through Day 29
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A SAE is defined as any serious adverse event that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, significant medical events that may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed before.
Time Frame: Up to Day 29
Population: Safety Population consisted of all randomized participants who were exposed to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 8 | 22
Participants
  All AEs | 0 | 3
  SAEs | 0 | 0

2. Primary Outcome: Part A: Number of Participants With Adverse Events of Special Interest (AESI) Through Day 29
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. AESIs were infusion-related reactions (IRR) including hypersensitivity, events related to antibody-dependent enhancement, and events related to immunogenicity.
Time Frame: Up to Day 29
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 8 | 22
Participants
  IRR including hypersensitivity | 0 | 0
  Events related to antibody-dependent enhancement | 0 | 0
  Events related to immunogenicity | 0 | 0

3. Primary Outcome: Part A: Number of Participants With Worst-case Post Baseline Abnormal Electrocardiogram (ECG) Findings Through Day 29
Description: Twelve-lead ECGs were recorded with the participant in a semi-supine position after being at rest for at least 10 minutes using an ECG machine. Clinically significant abnormal findings were determined as per clinical judgement by the investigator. Number of participants with worst-case clinically significant and not clinically significant abnormal ECG findings have been presented.
Time Frame: Up to Day 29
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 8 | 22
Participants
  Abnormal-Clinically significant | 0 | 0
  Abnormal-Not Clinically significant | 6 | 17

4. Primary Outcome: Part A: Number of Participants With Disease Progression Events (Disease-Related Events) Through Day 29
Description: AEs related to expected progression, signs, or symptoms of COVID-19, unless more severe than expected for the participant's current clinical status and medical history, and considered to be not causally-related to the study agent or study procedures by the Investigator, were reported as a Disease-Related Events (DRE).
Time Frame: Up to Day 29
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 8 | 22
Participants | 0 | 0

5. Primary Outcome: Part B: Mean Area Under the Curve (AUC) of Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Viral Load From Day 1 to Day 8 (AUCD1-8)
Description: AUC of SARS-CoV-2 viral load was measured by Quantitative reverse transcriptase polymerase chain reaction (qRT-PCR) from Day 1 to Day 8 in nasopharyngeal (NP) swab samples. Analysis was performed using an Analysis of covariance (ANCOVA) model with covariates of treatment and Baseline logarithm (base 10) viral load.
Time Frame: Day 1 to Day 8
Population: Viral Pharmacodynamic Population consisted of all participants in the Safety Population who had a Baseline (Day 1) quantifiable viral load as assessed using qRT-PCR from NP swabs. Only those participants with data available at the specified time points without missing covariate information were analyzed.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Day*log10 copies per (/) milliliter (mL)
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 64 | 65
Day*log10 copies per (/) milliliter (mL) | 24.40 [23.53 to 25.31] | 25.28 [24.38 to 26.21]
Statistical Analysis 1: Comparison: Part B- Sotrovimab Gen2: 500 mg IV vs Part B- Sotrovimab Gen2: 500 mg IM; Test type: Other; Ratio of geometric least squares mean = 1.04, 90% CI 2-sided [0.98 to 1.09] — Analysis was performed using an Analysis of covariance (ANCOVA) model with covariates of treatment and Baseline logarithm (base 10) viral load

6. Primary Outcome: Part C: Mean AUC of SARS-CoV-2 Viral Load From Day 1 to Day 8 (AUCD1-8)
Description: AUC of SARS-CoV-2 viral load was measured by qRT-PCR from Day 1 to Day 8 in NP swab samples. Analysis was performed using an ANCOVA model with covariates of treatment, and Baseline logarithm (base10) viral load and randomization stratification factor (prior exposure to an authorized or approved SARS-CoV-2 vaccine).
Time Frame: Day 1 to Day 8
Population: Viral Pharmacodynamic Population. Only those participants with data available at the specified time points without missing covariate information were analyzed.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Day*log10 copies/mL
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 55 | 62
Day*log10 copies/mL | 26.20 [24.68 to 27.81] | 26.72 [25.26 to 28.27]
Statistical Analysis 1: Comparison: Part C- Sotrovimab Gen2: 500 mg IV vs Part C- Sotrovimab Gen2: 250 mg IM; Test type: Other; Ratio of geometric least squares mean = 1.02, 90% CI 2-sided [0.94 to 1.11] — Analysis was performed using an ANCOVA model with covariates of treatment, and Baseline logarithm (base10) viral load and randomization stratification factor (prior exposure to an authorized or approved SARS-CoV-2 vaccine)

7. Secondary Outcome: Part A: Number of Participants With Non-Serious AEs Through Week 12
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Adverse events which were not Serious were considered as Non-Serious adverse events.
Time Frame: Up to Week 12
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 8 | 22
Participants | 0 | 0

8. Secondary Outcome: Part A: Number of Participants With SAEs Through Week 24
Description: A SAE is defined as any serious adverse event that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, significant medical events that may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed before.
Time Frame: Up to Week 24
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 8 | 22
Participants | 0 | 0

9. Secondary Outcome: Part A: Number of Participants With AESI Through Week 24
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. AESIs are infusion-related reactions (IRR) including hypersensitivity, events related to antibody-dependent enhancement, and events related to immunogenicity.
Time Frame: Up to Week 24
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 8 | 22
Participants
  IRR including hypersensitivity | 0 | 0
  Events related to antibody-dependent enhancement | 0 | 0
  Events related to immunogenicity | 0 | 0

10. Secondary Outcome: Part A: Number of Participants With Abnormal ECG Findings at Indicated Time Points
Description: Twelve-lead ECGs were recorded with the participant in a semi-supine position after being at rest for at least 10 minutes using an ECG machine. Clinically significant abnormal findings were determined as per clinical judgement by the investigator. Number of participants with clinically significant (CS) and not clinically significant (NCS) abnormal ECG findings have been presented.
Time Frame: Days 1, 5, 11 and 85 (Week 12)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 8 | 22
Participants
  Day 1: Abnormal-CS, n=7,22: number analyzed (Participants) | 7 | 22
  Day 1: Abnormal-CS, n=7,22 | 0 | 0
  Day 1:Abnormal-NCS, n=7,22: number analyzed (Participants) | 7 | 22
  Day 1:Abnormal-NCS, n=7,22 | 4 | 13
  Day 5: Abnormal-CS, n=7,21: number analyzed (Participants) | 7 | 21
  Day 5: Abnormal-CS, n=7,21 | 0 | 0
  Day 5:Abnormal-NCS, n=7,21: number analyzed (Participants) | 7 | 21
  Day 5:Abnormal-NCS, n=7,21 | 5 | 10
  Day 11: Abnormal-CS, n=8,22 | 0 | 0
  Day 11:Abnormal-NCS,n=8,22 | 5 | 12
  Day 85 (Week 12): Abnormal-CS, n=8,22 | 0 | 0
  Day 85 (Week 12):Abnormal-NCS,n=8,22 | 6 | 10

11. Secondary Outcome: Part A: Number of Participants With Disease Progression Events (Disease-Related Events) Through Week 24
Description: as for outcome 4
Time Frame: Up to Week 24
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 8 | 22
Participants | 0 | 0

12. Secondary Outcome: Part B: Number of Participants With All AEs and SAEs Through Day 29
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A SAE is defined as any serious adverse event that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, significant medical events that may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed before. Adverse events include both Serious and Other Adverse Events.
Time Frame: Up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 84 | 82
Participants
  All AEs | 8 | 17
  SAEs | 1 | 2

13. Secondary Outcome: Part B: Number of Participants With AESI Through Day 29
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. AESIs were infusion/injection-related reactions (IRR) including hypersensitivity; injection site reactions (ISRs); events related to antibody-dependent enhancement; events related to immunogenicity.
Time Frame: Up to Day 29
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 84 | 82
Participants
  IRR including hypersensitivity | 0 | 1
  Injection site reactions | 0 | 10
  Events related to antibody-dependent enhancement | 0 | 0
  Events related to immunogenicity | 0 | 0

14. Secondary Outcome: Part B: Number of Participants With Worst-case Post Baseline Abnormal ECG Findings Through Day 29
Description: as for outcome 3
Time Frame: Up to Day 29
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 84 | 82
Participants
  Abnormal-Clinically significant | 1 | 1
  Abnormal-Not Clinically significant | 43 | 39

15. Secondary Outcome: Part B: Number of Participants With Disease Progression Events (Disease-Related Events) Through Day 29
Description: as for outcome 4
Time Frame: Up to Day 29
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 84 | 82
Participants | 0 | 3

16. Secondary Outcome: Part C: Number of Participants With All AEs and SAEs Through Day 29
Description: as for outcome 12
Time Frame: Up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 79 | 78
Participants
  All AEs | 10 | 13
  SAEs | 1 | 3

17. Secondary Outcome: Part C: Number of Participants With AESI Through Day 29
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. AESIs were infusion/injection-related reactions (IRR) including hypersensitivity reactions; injection site reactions (ISRs); events related to antibody-dependent enhancement, and events related to immunogenicity.
Time Frame: Up to Day 29
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 79 | 78
Participants
  IRR including hypersensitivity | 0 | 0
  Injection site reactions | 0 | 4
  Events related to antibody-dependent enhancement | 0 | 0
  Events related to immunogenicity | 0 | 0

18. Secondary Outcome: Part C: Number of Participants With Worst-case Post Baseline Abnormal ECG Findings Through Day 29
Description: as for outcome 3
Time Frame: Up to Day 29
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 79 | 78
Participants
  Abnormal-Clinically significant | 0 | 0
  Abnormal-Not Clinically significant | 38 | 37

19. Secondary Outcome: Part C: Number of Participants With Disease Progression Events (Disease-Related Events) Through Day 29
Description: as for outcome 4
Time Frame: Up to Day 29
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 79 | 78
Participants | 0 | 0

20. Secondary Outcome: Part B: Number of Participants With Non-Serious AEs Through Week 12
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Time Frame: Up to Week 12
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 84 | 82
Participants | 8 | 20

21. Secondary Outcome: Part B: Number of Participants With SAEs Through Week 36
Description: as for outcome 8
Time Frame: Up to Week 36
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 84 | 82
Participants | 1 | 2

22. Secondary Outcome: Part B: Number of Participants With AESI Through Week 36
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. AESIs are infusion/injection-related reactions (IRR) including hypersensitivity reactions; injection site reactions (ISRs); events related to antibody-dependent enhancement, and events related to immunogenicity.
Time Frame: up to Week 36
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 84 | 82
Participants
  IRR including hypersensitivity reaction | 0 | 1
  Injection site reactions | 0 | 10
  Events related to antibody-dependent enhancement | 0 | 0
  Events related to immunogenicity | 0 | 0

23. Secondary Outcome: Part B: Number of Participants With Abnormal ECG Findings at Indicated Time Points
Description: as for outcome 10
Time Frame: Days 1, 5, 11 and 85 (Week 12)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 84 | 82
Participants
  Day 1: Abnormal-CS, n=84,82 | 1 | 0
  Day 1:Abnormal-NCS, n=84,82 | 33 | 31
  Day 5: Abnormal-CS, n=80,78: number analyzed (Participants) | 80 | 78
  Day 5: Abnormal-CS, n=80,78 | 0 | 1
  Day 5:Abnormal-NCS, n=80,78: number analyzed (Participants) | 80 | 78
  Day 5:Abnormal-NCS, n=80,78 | 28 | 24
  Day 11: Abnormal-CS, n=82,78: number analyzed (Participants) | 82 | 78
  Day 11: Abnormal-CS, n=82,78 | 0 | 0
  Day 11:Abnormal-NCS,n=82,78: number analyzed (Participants) | 82 | 78
  Day 11:Abnormal-NCS,n=82,78 | 20 | 24
  Day 85 (Week 12): Abnormal-CS, n=78,79: number analyzed (Participants) | 78 | 79
  Day 85 (Week 12): Abnormal-CS, n=78,79 | 0 | 0
  Day 85 (Week 12):Abnormal-NCS,n=78,79: number analyzed (Participants) | 78 | 79
  Day 85 (Week 12):Abnormal-NCS,n=78,79 | 24 | 20

24. Secondary Outcome: Part B: Number of Participants With Disease Progression Events Through Week 36
Description: as for outcome 4
Time Frame: Up to Week 36
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 84 | 82
Participants | 2 | 3

25. Secondary Outcome: Part C: Number of Participants With Non-Serious AEs Through Week 12
Description: as for outcome 20
Time Frame: Up to Week 12
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 79 | 78
Participants | 16 | 16

26. Secondary Outcome: Part C: Number of Participants With SAEs Through Week 36
Description: as for outcome 8
Time Frame: Up to Week 36
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 79 | 78
Participants | 2 | 3

27. Secondary Outcome: Part C: Number of Participants With AESI Through Week 36
Description: as for outcome 22
Time Frame: Up to Week 36
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 79 | 78
Participants
  IRR including hypersensitivity | 0 | 0
  Injection site reactions | 0 | 4
  Events related to antibody-dependent enhancement | 0 | 0
  Events related to immunogenicity | 0 | 0

28. Secondary Outcome: Part C: Number of Participants With Abnormal ECG Findings at Indicated Time Points
Description: as for outcome 10
Time Frame: Days 1, 5, 11 and 85 (Week 12)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 79 | 78
Participants
  Day 1: Abnormal-CS, n=79,78 | 0 | 0
  Day 1:Abnormal-NCS, n=79,78 | 29 | 28
  Day 5: Abnormal-CS, n=76,74: number analyzed (Participants) | 76 | 74
  Day 5: Abnormal-CS, n=76,74 | 0 | 0
  Day 5:Abnormal-NCS, n=76,74: number analyzed (Participants) | 76 | 74
  Day 5:Abnormal-NCS, n=76,74 | 25 | 23
  Day 11: Abnormal-CS, n=72,76: number analyzed (Participants) | 72 | 76
  Day 11: Abnormal-CS, n=72,76 | 0 | 0
  Day 11:Abnormal-NCS,n=72,76: number analyzed (Participants) | 72 | 76
  Day 11:Abnormal-NCS,n=72,76 | 21 | 23
  Day 85 (Week 12): Abnormal-CS, n=73,77: number analyzed (Participants) | 73 | 77
  Day 85 (Week 12): Abnormal-CS, n=73,77 | 0 | 0
  Day 85 (Week 12):Abnormal-NCS,n=73,77: number analyzed (Participants) | 73 | 77
  Day 85 (Week 12):Abnormal-NCS,n=73,77 | 20 | 23

29. Secondary Outcome: Part C: Number of Participants With Disease Progression Events Through Week 36
Description: as for outcome 4
Time Frame: Up to Week 36
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 79 | 78
Participants | 1 | 4

30. Secondary Outcome: Part A: Change From Baseline in SARS-CoV-2 Saliva and Nasal Mid-Turbinate Viral Load
Description: SARS-CoV-2 viral load was based on saliva and nasal mid-turbinate swab samples and was measured by qRT-PCR. Baseline log10 viral load was defined as the non-missing assessment taken at Day 1 excluding the NEG and <2.08 results. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline, Days 2, 5, 8, 11, 15, 22 and 29
Population: Virology Population consisted of all participants in the Safety Population with a central lab confirmed quantifiable nasal mid-turbinate and/or saliva swab at Baseline. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 6 | 16
Log10 copies/mL
  Day 2: Saliva, n=4,11: number analyzed (Participants) | 4 | 11
  Day 2: Saliva, n=4,11 | -0.270 (0.4290) | -1.114 (0.9201)
  Day 5: Saliva, n=3,11: number analyzed (Participants) | 3 | 11
  Day 5: Saliva, n=3,11 | -0.780 (0.3404) | -2.620 (1.0199)
  Day 8: Saliva, n=3,11: number analyzed (Participants) | 3 | 11
  Day 8: Saliva, n=3,11 | -0.507 (0.5689) | -2.605 (1.4982)
  Day 11: Saliva, n=4,10: number analyzed (Participants) | 4 | 10
  Day 11: Saliva, n=4,10 | -1.043 (0.5940) | -2.881 (1.3963)
  Day 15: Saliva, n=4,11: number analyzed (Participants) | 4 | 11
  Day 15: Saliva, n=4,11 | -0.610 (1.3444) | -3.179 (1.2132)
  Day 22: Saliva, n=4,11: number analyzed (Participants) | 4 | 11
  Day 22: Saliva, n=4,11 | -1.043 (0.5940) | -3.284 (1.3210)
  Day 29: Saliva, n=4,11: number analyzed (Participants) | 4 | 11
  Day 29: Saliva, n=4,11 | -1.043 (0.5940) | -3.223 (1.3123)
  Day 2: Nasal mid-turbinate, n=5,16: number analyzed (Participants) | 5 | 16
  Day 2: Nasal mid-turbinate, n=5,16 | -1.252 (0.9726) | -1.006 (1.2277)
  Day 5: Nasal mid-turbinate, n=4,16: number analyzed (Participants) | 4 | 16
  Day 5: Nasal mid-turbinate, n=4,16 | -1.755 (1.1230) | -2.111 (1.2100)
  Day 8: Nasal mid-turbinate, n=4,16: number analyzed (Participants) | 4 | 16
  Day 8: Nasal mid-turbinate, n=4,16 | -1.705 (0.7839) | -2.703 (1.7842)
  Day 11: Nasal mid-turbinate, n=5,16: number analyzed (Participants) | 5 | 16
  Day 11: Nasal mid-turbinate, n=5,16 | -2.810 (1.3363) | -2.923 (1.5656)
  Day 15: Nasal mid-turbinate, n=5,16: number analyzed (Participants) | 5 | 16
  Day 15: Nasal mid-turbinate, n=5,16 | -2.490 (1.3243) | -3.445 (1.7103)
  Day 22: Nasal mid-turbinate, n=5,16: number analyzed (Participants) | 5 | 16
  Day 22: Nasal mid-turbinate, n=5,16 | -2.668 (1.2826) | -3.873 (1.9434)
  Day 29: Nasal mid-turbinate, n=5,16: number analyzed (Participants) | 5 | 16
  Day 29: Nasal mid-turbinate, n=5,16 | -2.810 (1.3363) | -3.752 (1.8030)

31. Secondary Outcome: Part B: Change From Baseline in Viral Load as Measured by qRT-PCR From Nasopharyngeal Swab Samples
Description: Viral load was based on nasopharyngeal swab samples and was measured by qRT-PCR. Baseline log10 viral load was defined as the non-missing assessment taken at Day 1 excluding the "NEG" and "<2.08" results. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline, Days 2, 3, 5, 8, 11, 15, 22 and 29
Population: Viral Pharmacodynamic Population consisted of all participants in the Safety Population who had a Baseline (Day 1) quantifiable viral load as assessed using qRT-PCR from NP swabs. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 66 | 68
Log10 copies/mL
  Day 2: n=63,68: number analyzed (Participants) | 63 | 68
  Day 2: n=63,68 | -1.146 (1.1558) | -0.611 (1.1518)
  Day 3: n=63,66: number analyzed (Participants) | 63 | 66
  Day 3: n=63,66 | -1.438 (1.2033) | -1.306 (1.3132)
  Day 5: n=62,64: number analyzed (Participants) | 62 | 64
  Day 5: n=62,64 | -2.578 (1.2480) | -2.352 (1.1655)
  Day 8: n=64,64: number analyzed (Participants) | 64 | 64
  Day 8: n=64,64 | -3.069 (1.4553) | -3.254 (1.4193)
  Day 11: n=62,63: number analyzed (Participants) | 62 | 63
  Day 11: n=62,63 | -3.522 (1.7148) | -3.574 (1.4907)
  Day 15: n=62,66: number analyzed (Participants) | 62 | 66
  Day 15: n=62,66 | -3.705 (1.7443) | -3.733 (1.5525)
  Day 22: n=64,66: number analyzed (Participants) | 64 | 66
  Day 22: n=64,66 | -3.831 (1.7994) | -3.778 (1.7476)
  Day 29: n=62,64: number analyzed (Participants) | 62 | 64
  Day 29: n=62,64 | -3.933 (1.8253) | -3.857 (1.7455)

32. Secondary Outcome: Part C: Change From Baseline in Viral Load as Measured by qRT-PCR From Nasopharyngeal Swab Samples
Description: as for outcome 31
Time Frame: Baseline, Days 2, 3, 5, 8, 11, 15, 22 and 29
Population: Viral Pharmacodynamic Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Log10 copies per milliliter
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 61 | 66
Log10 copies per milliliter
  Day 2: n=59,64: number analyzed (Participants) | 59 | 64
  Day 2: n=59,64 | -0.429 (1.3835) | -0.519 (1.3273)
  Day 3: n=50,57: number analyzed (Participants) | 50 | 57
  Day 3: n=50,57 | -0.905 (1.5202) | -1.123 (1.6172)
  Day 5: n=57,62: number analyzed (Participants) | 57 | 62
  Day 5: n=57,62 | -2.076 (1.9648) | -1.967 (2.0218)
  Day 8: n=55,62: number analyzed (Participants) | 55 | 62
  Day 8: n=55,62 | -3.122 (1.8234) | -3.180 (1.8324)
  Day 11: n=52,61: number analyzed (Participants) | 52 | 61
  Day 11: n=52,61 | -3.617 (1.6870) | -3.738 (1.8168)
  Day 15: n=50,61: number analyzed (Participants) | 50 | 61
  Day 15: n=50,61 | -3.719 (1.8248) | -3.836 (1.8148)
  Day 22: n=55,65: number analyzed (Participants) | 55 | 65
  Day 22: n=55,65 | -3.693 (1.7647) | -3.956 (1.7492)
  Day 29: n=56,63: number analyzed (Participants) | 56 | 63
  Day 29: n=56,63 | -3.761 (1.8167) | -3.963 (1.7189)

33. Secondary Outcome: Part B: Percentage of Participants With Undetectable Viral Load
Description: Viral load was measured by qRT-PCR from nasopharyngeal swab samples. Viral load (log10 copies/mL) values recorded as negative were considered as undetectable viral load. Percentage of participants with undetectable viral load have been presented. Percentage values are rounded off.
Time Frame: Days 2, 3, 5, 8, 11, 15, 22 and 29
Population: Viral Pharmacodynamic Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Number; unit: Percentage of participants
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 66 | 68
Percentage of participants
  Day 2: n=63,68: number analyzed (Participants) | 63 | 68
  Day 2: n=63,68 | 10 | 4
  Day 3: n=63,66: number analyzed (Participants) | 63 | 66
  Day 3: n=63,66 | 11 | 9
  Day 5: n=62,64: number analyzed (Participants) | 62 | 64
  Day 5: n=62,64 | 23 | 27
  Day 8: n=64,64: number analyzed (Participants) | 64 | 64
  Day 8: n=64,64 | 34 | 38
  Day 11: n=62,63: number analyzed (Participants) | 62 | 63
  Day 11: n=62,63 | 58 | 51
  Day 15: n=62,66: number analyzed (Participants) | 62 | 66
  Day 15: n=62,66 | 61 | 73
  Day 22: n=64,66: number analyzed (Participants) | 64 | 66
  Day 22: n=64,66 | 73 | 74
  Day 29: n=62,64: number analyzed (Participants) | 62 | 64
  Day 29: n=62,64 | 81 | 84

34. Secondary Outcome: Part C: Percentage of Participants With Undetectable Viral Load
Description: as for outcome 33
Time Frame: Days 2, 3, 5, 8, 11, 15, 22 and 29
Population: as for outcome 33
Measure: Number; unit: Percentage of participants
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 61 | 66
Percentage of participants
  Day 2: n=59,64: number analyzed (Participants) | 59 | 64
  Day 2: n=59,64 | 10 | 5
  Day 3: n=50,57: number analyzed (Participants) | 50 | 57
  Day 3: n=50,57 | 10 | 14
  Day 5: n=57,62: number analyzed (Participants) | 57 | 62
  Day 5: n=57,62 | 28 | 16
  Day 8: n=55,62: number analyzed (Participants) | 55 | 62
  Day 8: n=55,62 | 42 | 39
  Day 11: n=52,61: number analyzed (Participants) | 52 | 61
  Day 11: n=52,61 | 63 | 72
  Day 15: n=50,61: number analyzed (Participants) | 50 | 61
  Day 15: n=50,61 | 82 | 80
  Day 22: n=55,65: number analyzed (Participants) | 55 | 65
  Day 22: n=55,65 | 80 | 88
  Day 29: n=56,63: number analyzed (Participants) | 56 | 63
  Day 29: n=56,63 | 88 | 86

35. Secondary Outcome: Part B: Mean AUC of SARS-CoV-2 Viral Load From Day 1 to Day 5 (AUCD1-5)
Description: AUC of SARS-CoV-2 viral load was measured by qRT-PCR from Day 1 to Day 5. Analysis was performed using an ANCOVA model with covariates of treatment and Baseline logarithm (base 10) viral load.
Time Frame: Day 1 to Day 5
Population: as for outcome 6
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Day*log10 copies/mL
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 63 | 65
Day*log10 copies/mL | 16.14 [15.53 to 16.77] | 16.97 [16.34 to 17.62]
Statistical Analysis 1: Comparison: Part B- Sotrovimab Gen2: 500 mg IV vs Part B- Sotrovimab Gen2: 500 mg IM; Test type: Other; Ratio of geometric least squares mean = 1.05, 90% CI 2-sided [1.00 to 1.11] — Analysis was performed using an ANCOVA model with covariates of treatment and Baseline logarithm (base 10) viral load

36. Secondary Outcome: Part B: Mean Area Under the Curve (AUC) of SARS-CoV-2 Viral Load From Day 1 to Day 11 (AUCD1-11)
Description: AUC of SARS-CoV-2 viral load was measured by qRT-PCR from Day 1 to Day 11. Analysis was performed using an ANCOVA model with covariates of treatment and Baseline logarithm (base 10) viral load.
Time Frame: Day 1 to Day 11
Population: as for outcome 6
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Day*log10 copies/mL
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 64 | 65
Day*log10 copies/mL | 31.69 [30.60 to 32.82] | 32.39 [31.28 to 33.53]
Statistical Analysis 1: Comparison: Part B- Sotrovimab Gen2: 500 mg IV vs Part B- Sotrovimab Gen2: 500 mg IM; Test type: Other; Ratio of geometric least squares mean = 1.02, 90% CI 2-sided [0.97 to 1.07] — Analysis was performed using an ANCOVA model with covariates of treatment and Baseline logarithm (base 10) viral load

37. Secondary Outcome: Part C: Mean AUC of SARS-CoV-2 Viral Load From Day 1 to Day 5 (AUCD1-5)
Description: AUC of SARS-CoV-2 viral load was measured by qRT-PCR from Day 1 to Day 5. Analysis was performed using an ANCOVA model with covariates of treatment, Baseline logarithm (base 10) viral load and randomization stratification factor (prior exposure to an authorized or approved SARS-CoV-2 vaccine).
Time Frame: Day 1 to Day 5
Population: as for outcome 6
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Day*log10 copies/mL
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 57 | 63
Day*log10 copies/mL | 17.42 [16.49 to 18.41] | 17.56 [16.66 to 18.51]
Statistical Analysis 1: Comparison: Part C- Sotrovimab Gen2: 500 mg IV vs Part C- Sotrovimab Gen2: 250 mg IM; Test type: Other; Ratio of geometric least squares mean = 1.01, 90% CI 2-sided [0.93 to 1.09] — Analysis was performed using an ANCOVA model with covariates of treatment, Baseline logarithm (base 10) viral load and randomization stratification factor (prior exposure to an authorized or approved SARS-CoV-2 vaccine)

38. Secondary Outcome: Part C: Mean Area Under the Curve (AUC) of SARS-CoV-2 Viral Load From Day 1 to Day 11 (AUCD1-11)
Description: AUC of SARS-CoV-2 viral load was measured by qRT-PCR from Day 1 to Day 11. Analysis was performed using an ANCOVA model with covariates of treatment, Baseline logarithm (base 10) viral load and randomization stratification factor (prior exposure to an authorized or approved SARS-CoV-2 vaccine).
Time Frame: Day 1 to Day 11
Population: as for outcome 6
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Day*log10 copies/mL
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 53 | 62
Day*log10 copies/mL | 33.02 [31.17 to 34.97] | 33.63 [31.89 to 35.47]
Statistical Analysis 1: Comparison: Part C- Sotrovimab Gen2: 500 mg IV vs Part C- Sotrovimab Gen2: 250 mg IM; Test type: Other; Ratio of geometric least squares mean = 1.02, 90% CI 2-sided [0.94 to 1.10] — [estimate comment as in outcome 37, analysis 1]

39. Secondary Outcome: Part B: Percentage of Participants With a Persistently High Viral Load at Day 8
Description: Percentage of participants with a persistently high viral load were categorized as >=4.1 log10 copies/mL and <4.1 log10 copies/mL. Percentage of participants with a persistently high viral load at Day 8 was assessed via qRT-PCR in nasopharyngeal swab samples. Percentage of participants with a persistently high viral load at Day 8 has been presented. Percentage values are rounded off.
Time Frame: Day 8
Population: Viral Pharmacodynamic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 64 | 64
Percentage of participants
  >=4.1 log 10 copies/mL | 17 | 11
  <4.1 log 10 copies/mL | 83 | 89

40. Secondary Outcome: Part C: Percentage of Participants With a Persistently High Viral Load at Day 8
Description: as for outcome 39
Time Frame: Day 8
Population: as for outcome 39
Measure: Number; unit: Percentage of participants
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 55 | 62
Percentage of participants
  >=4.1 log 10 copies/mL | 15 | 13
  <4.1 log 10 copies/mL | 85 | 87

41. Secondary Outcome: Part A: Maximum Observed Concentration (Cmax) of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion and at 1, 2, 6, and 8 hours following end of infusion; Days 2, 5, 8, 15, 29, 43, 57, 85, 141, and 169 (+/-12 days)
Population: Pharmacokinetic Population consisted of all participants in the Safety Population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values were considered as non-missing values). Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per mL
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 7 | 22
Microgram per mL | 147.1 (48.28) | 204.7 (77.61)

42. Secondary Outcome: Part B: Cmax of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per mL
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 6
Microgram per mL | 156.5 (40.80)

43. Secondary Outcome: Part B: Cmax of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Microgram per mL
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 11
Microgram per mL | 28.8 (15.66)

44. Secondary Outcome: Part C: Cmax of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per mL
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 5
Microgram per mL | 137.4 (32.97)

45. Secondary Outcome: Part C: Cmax of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per mL
Arm/Group | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 7
Microgram per mL | 11.1 (5.61)

46. Secondary Outcome: Part A: Concentration at Last Quantifiable Time-point (Clast) of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: as for outcome 41
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Microgram per mL
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 8 | 22
Microgram per mL | 6.9 (2.16) | 8.1 (2.17)

47. Secondary Outcome: Part B: Clast of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Microgram per mL
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 11
Microgram per mL | 7.0 (2.48)

48. Secondary Outcome: Part B: Clast of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Microgram per mL
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 11
Microgram per mL | 7.9 (7.65)

49. Secondary Outcome: Part C: Clast of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Microgram per mL
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 10
Microgram per mL | 10.5 (12.59)

50. Secondary Outcome: Part C: Clast of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Microgram per mL
Arm/Group | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 10
Microgram per mL | 2.6 (1.73)

51. Secondary Outcome: Part A: Time to Reach Cmax (Tmax) of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: as for outcome 41
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Day
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 7 | 22
Day | 0.042 [0.04 to 0.38] | 0.042 [0.04 to 0.38]

52. Secondary Outcome: Part B: Tmax of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Day
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 6
Day | 0.026 [0.01 to 0.03]

53. Secondary Outcome: Part B: Tmax of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Day
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 11
Day | 6.878 [3.68 to 56.66]

54. Secondary Outcome: Part C: Tmax of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Day
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 5
Day | 0.014 [0.01 to 0.02]

55. Secondary Outcome: Part C: Tmax of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Day
Arm/Group | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 7
Day | 27.866 [13.88 to 56.04]

56. Secondary Outcome: Part A: Time of the Last Quantifiable Concentration (Tlast) of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: as for outcome 41
Population: Pharmacokinetic Population. The time frame is beyond Day 169 as there was one PK sample collected outside of the protocol defined window of +/- 7 days that was included in the analysis (PK sample collected up to Day 169 +/- 12 days).
Measure: Median (Full Range); unit: Day
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 8 | 22
Day | 161.333 [160.89 to 174.95] | 162.248 [160.70 to 180.15]

57. Secondary Outcome: Part B: Tlast of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population. The upper value of the full range is outside of the time frame due to the protocol defined time point of Day 169+/-7 days.
Measure: Median (Full Range); unit: Day
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 11
Day | 167.715 [160.76 to 175.68]

58. Secondary Outcome: Part B: Tlast of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: as for outcome 57
Measure: Median (Full Range); unit: Day
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 11
Day | 167.670 [55.68 to 175.66]

59. Secondary Outcome: Part C: Tlast of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. The time frame is beyond Day 169 as there were a few PK samples collected outside of the protocol defined window of +/- 7 days that were included in the analysis (PK samples collected up to Day 169 +/- 18 days).
Measure: Median (Full Range); unit: Day
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 10
Day | 162.458 [27.79 to 185.75]

60. Secondary Outcome: Part C: Tlast of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: as for outcome 59
Measure: Median (Full Range); unit: Day
Arm/Group | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 10
Day | 168.912 [160.97 to 180.83]

61. Secondary Outcome: Part A: AUC From Day 1 to 29 (AUCD1-29) of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion and at 1, 2, 6, and 8 hours following end of infusion; Days 2, 5, 8, 15, 29
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 8 | 22
Day*microgram/mL | 1355.2 (392.56) | 1738.8 (308.31)

62. Secondary Outcome: Part B: AUCD1-29 of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29 (+/-2 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 11
Day*microgram/mL | 1442.9 (296.96)

63. Secondary Outcome: Part B: AUCD1-29 of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29 (+/-2 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 11
Day*microgram/mL | 686.9 (376.78)

64. Secondary Outcome: Part C: AUCD1-29 of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29 (+/-2 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 10
Day*microgram/mL | 1405.4 (528.26)

65. Secondary Outcome: Part C: AUCD1-29 of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29 (+/-2 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 10
Day*microgram/mL | 327.1 (242.84)

66. Secondary Outcome: Part A: Area Under the Serum Concentration-time Curve Extrapolated From Zero to Infinity (AUC[0-inf]) of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: as for outcome 41
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 7 | 21
Day*microgram/mL | 3982.7 (1289.19) | 5238.4 (966.33)

67. Secondary Outcome: Part B: AUC(0-inf) of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 11
Day*microgram/mL | 4449.3 (1123.41)

68. Secondary Outcome: Part B: AUC(0-inf) of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 8
Day*microgram/mL | 3194.4 (1617.36)

69. Secondary Outcome: Part C: AUC(0-inf) of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 9
Day*microgram/mL | 4255.3 (1369.36)

70. Secondary Outcome: Part C: AUC(0-inf) of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 8
Day*microgram/mL | 1441.0 (985.65)

71. Secondary Outcome: Part A: Area Under the Curve From the Time of Dosing to the Time of the Last Measurable (Positive) Concentration (AUClast) of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: as for outcome 41
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 8 | 22
Day*microgram/mL | 3456.5 (1086.56) | 4528.5 (826.89)

72. Secondary Outcome: Part B: AUClast of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 11
Day*microgram/mL | 3848.5 (899.51)

73. Secondary Outcome: Part B: AUClast of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 11
Day*microgram/mL | 2446.5 (1249.20)

74. Secondary Outcome: Part C: AUClast of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 10
Day*microgram/mL | 3492.6 (1257.27)

75. Secondary Outcome: Part C: AUClast of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Day*microgram/mL
Arm/Group | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 10
Day*microgram/mL | 1185.8 (763.78)

76. Secondary Outcome: Part A: Percentage of AUC(Infinity) Obtained by Extrapolation (%AUCexp) for VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: as for outcome 41
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of AUCexp
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 7 | 21
Percentage of AUCexp | 14.9 (2.81) | 12.6 (3.42)

77. Secondary Outcome: Part B: %AUCexp of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Percentage of AUCexp
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 11
Percentage of AUCexp | 13.1 (2.92)

78. Secondary Outcome: Part B: %AUCexp of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of AUCexp
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 8
Percentage of AUCexp | 15.0 (2.35)

79. Secondary Outcome: Part C: %AUCexp of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of AUCexp
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 9
Percentage of AUCexp | 13.6 (4.29)

80. Secondary Outcome: Part C: %AUCexp of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of AUCexp
Arm/Group | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 8
Percentage of AUCexp | 15.0 (2.11)

81. Secondary Outcome: Part A: Terminal Elimination Half-life (t1/2) of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: as for outcome 41
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Day
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 7 | 21
Day | 63.196 [53.98 to 68.09] | 55.547 [42.34 to 72.09]

82. Secondary Outcome: Part B: t1/2 of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Day
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 11
Day | 55.735 [47.33 to 66.86]

83. Secondary Outcome: Part B: t1/2 of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Day
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 8
Day | 59.347 [51.95 to 65.83]

84. Secondary Outcome: Part C: t1/2 of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Day
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 9
Day | 60.938 [42.96 to 70.84]

85. Secondary Outcome: Part C: t1/2 of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Day
Arm/Group | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 8
Day | 61.867 [46.84 to 68.43]

86. Secondary Outcome: Part A: Apparent Volume of Distribution During the Elimination Phase Following Intravascular Administrtion (Vz) of VIR-7831
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: as for outcome 41
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 7 | 21
Liter | 12.40 (4.625) | 7.88 (1.374)

87. Secondary Outcome: Part B: Vz of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 11
Liter | 9.97 (2.865)

88. Secondary Outcome: Part B: Apparent Volume of Distribution During the Elimination Phase Following Extravascular Administration (Vz/F) of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 8
Liter | 18.14 (12.752)

89. Secondary Outcome: Part C: Vz of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 9
Liter | 10.93 (3.574)

90. Secondary Outcome: Part C: Vz/F of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 8
Liter | 20.24 (10.205)

91. Secondary Outcome: Part A: Apparent Volume of Distribution at Steady State (Vss) of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: as for outcome 41
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 7 | 21
Liter | 11.42 (4.110) | 7.47 (1.232)

92. Secondary Outcome: Part B: Vss of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 11
Liter | 9.41 (2.514)

93. Secondary Outcome: Part C: Vss of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 9
Liter | 10.61 (3.973)

94. Secondary Outcome: Part A: Clearance (CL) of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: as for outcome 41
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter per day
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 7 | 21
Milliliter per day | 136.8 (42.88) | 98.7 (18.62)

95. Secondary Outcome: Part B: CL of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Milliliter per day
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 11
Milliliter per day | 120.3 (35.96)

96. Secondary Outcome: Part B: Apparent Clearance (CL/F) of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-7 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter per day
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 8
Milliliter per day | 216.2 (162.28)

97. Secondary Outcome: Part C: CL of VIR-7831 After IV Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose, end of infusion; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter per day
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 9
Milliliter per day | 130.5 (47.83)

98. Secondary Outcome: Part C: CL/F of VIR-7831 After IM Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter per day
Arm/Group | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 8
Milliliter per day | 237.8 (125.67)

99. Secondary Outcome: Dose-normalized Least Square Geometric Mean Ratio of AUCinf for VIR-7831 Gen2 Between the Three Dose Levels (250 mg IM in Part C, 500 mg IM in Part B and 500 mg IV in Parts B and C)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab). Dose-normalized least square geometric mean ratio of AUCinf was derived based on collected assessments up to 169 (+/-7 days) for Part B- Sotrovimab Gen2: 500 mg IV arm, and up to 169 (+/-18 days) for Part C- Sotrovimab Gen2: 500 mg IV arm.
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed. Data from Parts B and C is presented in a single outcome to determine the absolute bioavailability (F) based on the loge transformed dose normalized AUCinf for the IV (500 mg), IM (500 mg), and IM (250 mg). Data for 500 mg IV arms with similar dosing strategies across Parts B and C is combined as pre-specified in reporting and analysis plan.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Day*microgram/mL
Groups:
- Sotrovimab Gen2: 500 mg IV (Parts B and C): Participants received Sotrovimab (VIR-7831) Gen2 500 mg IV infusion on Day 1 in Parts B and C.
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM | Part C- Sotrovimab Gen2: 250 mg IM | Sotrovimab Gen2: 500 mg IV (Parts B and C)
Number analyzed (Participants) | 8 | 8 | 20
Day*microgram/mL | 5.52 [4.25 to 7.16] | 4.86 [3.75 to 6.30] | 8.40 [7.12 to 9.90]
Statistical Analysis 1: Comparison: Part B- Sotrovimab Gen2: 500 mg IM vs Sotrovimab Gen2: 500 mg IV (Parts B and C); Test type: Other; Ratio of geometric least squares mean = 0.66, 90% CI 2-sided [0.48 to 0.89] — Drug bioavailability was analyzed using an ANCOVA model with treatment and weight at Baseline as covariates
Statistical Analysis 2: Comparison: Part C- Sotrovimab Gen2: 250 mg IM vs Sotrovimab Gen2: 500 mg IV (Parts B and C); Test type: Other; Ratio of geometric least squares mean = 0.58, 90% CI 2-sided [0.43 to 0.79] — Drug bioavailability was analyzed using an ANCOVA model with treatment and weight at Baseline as covariates

100. Secondary Outcome: Dose-normalized Least Square Geometric Mean Ratio of AUCinf for VIR-7831 Gen2 Between the Two IM Dose Levels (250 mg IM in Part C and 500 mg IM in Part B)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Day*microgram per milliliter
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 8 | 8
Day*microgram per milliliter | 5.56 [3.81 to 8.11] | 4.86 [3.33 to 7.09]
Statistical Analysis 1: Comparison: Part B- Sotrovimab Gen2: 500 mg IM vs Part C- Sotrovimab Gen2: 250 mg IM; Test type: Other; Ratio of geometric least squares mean = 1.14, 90% CI 2-sided [0.67 to 1.95] — Dose proportionality was analyzed using an ANOVA model with treatment (250mg, 500mg) as a covariate, for each parameter of interest

101. Secondary Outcome: Dose-normalized Least Square Geometric Mean Ratio of AUClast for VIR-7831 Gen2 Between the Two IM Dose Levels (250 mg IM in Part C and 500 mg IM in Part B)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Day*microgram per milliliter
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 11 | 10
Day*microgram per milliliter | 4.31 [3.21 to 5.77] | 4.05 [2.98 to 5.51]
Statistical Analysis 1: Comparison: Part B- Sotrovimab Gen2: 500 mg IM vs Part C- Sotrovimab Gen2: 250 mg IM; Test type: Other; Ratio of geometric least squares mean = 1.06, 90% CI 2-sided [0.69 to 1.62] — [estimate comment as in outcome 100, analysis 1]

102. Secondary Outcome: Dose-normalized Least Square Geometric Mean Ratio of AUCD1-D29 for VIR-7831 Gen2 Between the Two IM Dose Levels (250 mg IM in Part C and 500 mg IM in Part B)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29 (+/-2 days)
Population: Pharmacokinetic Population.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Day*microgram per milliliter
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 11 | 10
Day*microgram per milliliter | 1.17 [0.83 to 1.65] | 1.06 [0.74 to 1.51]
Statistical Analysis 1: Comparison: Part B- Sotrovimab Gen2: 500 mg IM vs Part C- Sotrovimab Gen2: 250 mg IM; Test type: Other; Ratio of geometric least squares mean = 1.11, 90% CI 2-sided [0.68 to 1.82] — [estimate comment as in outcome 100, analysis 1]

103. Secondary Outcome: Dose-normalized Least Square Geometric Mean Ratio of Cmax for VIR-7831 Gen2 Between the Two IM Dose Levels (250 mg IM in Part C and 500 mg IM in Part B)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of VIR-7831 (Sotrovimab).
Time Frame: Day 1: Pre-dose; Days 2, 3, 5, 8, 15, 29, 57, 85, 141, and 169 (+/-18 days)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Microgram per milliliter
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IM | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 11 | 7
Microgram per milliliter | 0.05 [0.04 to 0.07] | 0.04 [0.03 to 0.06]
Statistical Analysis 1: Comparison: Part B- Sotrovimab Gen2: 500 mg IM vs Part C- Sotrovimab Gen2: 250 mg IM; Test type: Other; Ratio of geometric least squares mean = 1.28, 90% CI 2-sided [0.77 to 2.12] — [estimate comment as in outcome 100, analysis 1]

104. Other Pre Specified Outcome: Part A: Number of Participants With Presence of SARS-CoV-2 Viral Resistance Mutants Against VIR-7831
Description: Number of participants with presence of SARS-CoV-2 viral resistance mutants against VIR-7831 was planned to be evaluated. The results for this outcome measure will never be posted.
Time Frame: Up to Day 28
Population: Safety Population. This was an other pre-specified outcome measure. The results for this outcome measure will never be posted.
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 0 | 0

105. Other Pre Specified Outcome: Part B: Number of Participants With Presence of SARS-CoV-2 Viral Resistance Mutants Against VIR-7831
Description: as for outcome 104
Time Frame: Up to Day 28
Population: as for outcome 104
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 0 | 0

106. Other Pre Specified Outcome: Part C: Number of Participants With Presence of SARS-CoV-2 Viral Resistance Mutants Against VIR-7831
Description: as for outcome 104
Time Frame: Up to Day 28
Population: as for outcome 104
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 0 | 0

107. Other Pre Specified Outcome: Part A: Number of Participants With Emergence of SARS-CoV-2 Viral Resistance Mutants Against VIR-7831
Description: Number of participants with emergence of SARS-CoV-2 viral resistance mutants against VIR-7831 was planned to be evaluated. The results for this outcome measure will never be posted.
Time Frame: Up to Day 28
Population: as for outcome 104
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 0 | 0

108. Other Pre Specified Outcome: Part B: Number of Participants With Emergence of SARS-CoV-2 Viral Resistance Mutants Against VIR-7831
Description: as for outcome 107
Time Frame: Up to Day 28
Population: as for outcome 104
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 0 | 0

109. Other Pre Specified Outcome: Part C: Number of Participants With Emergence of SARS-CoV-2 Viral Resistance Mutants Against VIR-7831
Description: as for outcome 107
Time Frame: Up to Day 28
Population: as for outcome 104
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 0 | 0

110. Other Pre Specified Outcome: Part A: Number of Participants With the Presence of Anti-VIR-7831 Antibody
Description: Number of participants with the presence of anti-VIR-7831 antibody was planned to be evaluated. The results for this outcome measure will never be posted.
Time Frame: Up to Week 24
Population: as for outcome 104
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 0 | 0

111. Other Pre Specified Outcome: Part B: Number of Participants With the Presence of Anti-VIR-7831 Antibody
Description: as for outcome 110
Time Frame: Up to Week 24
Population: as for outcome 104
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 0 | 0

112. Other Pre Specified Outcome: Part C: Number of Participants With the Presence of Anti-VIR-7831 Antibody
Description: as for outcome 110
Time Frame: Up to Week 24
Population: as for outcome 104
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 0 | 0

113. Other Pre Specified Outcome: Part A: Titers of Anti-drug Antibody to VIR-7831
Description: Serum samples were planned to be collected for the determination of anti-drug antibody using a validated electrochemiluminescent (ECL) immunoassay. The results for this outcome measure will never be posted.
Time Frame: Up to Week 24
Population: as for outcome 104
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 0 | 0

114. Other Pre Specified Outcome: Part B: Titers of Anti-drug Antibody to VIR-7831
Description: Serum samples were planned to be collected for the determination of anti-drug antibody using a validated ECL immunoassay. The results for this outcome measure will never be posted.
Time Frame: Up to Week 24
Population: as for outcome 104
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 0 | 0

115. Other Pre Specified Outcome: Part C: Titers of Anti-drug Antibody to VIR-7831
Description: as for outcome 114
Time Frame: Up to Week 24
Population: as for outcome 104
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 0 | 0

116. Other Pre Specified Outcome: Part A: Number of Participants With the Presence of Anti-nucleocapsid (Anti-N), Anti-spike (Anti-S) and Anti-Receptor Binding Domain (Anti-RBD) SARS-CoV-2 Antibodies at Baseline
Description: Number of participants with the presence of Anti-N, Anti-S and Anti-RBD SARS-CoV-2 antibodies were planned to be evaluated. The results for this outcome measure will never be posted.
Time Frame: Baseline (Day 1)
Population: as for outcome 104
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 0 | 0

117. Other Pre Specified Outcome: Part B: Number of Participants With the Presence of Anti-N, Anti-S and Anti-RBD SARS-CoV-2 Antibodies at Baseline
Description: as for outcome 116
Time Frame: Baseline (Day 1)
Population: as for outcome 104
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 0 | 0

118. Other Pre Specified Outcome: Part C: Number of Participants With the Presence of Anti-N, Anti-S and Anti-RBD SARS-CoV-2 Antibodies at Baseline
Description: as for outcome 116
Time Frame: Baseline (Day 1)
Population: as for outcome 104
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 0 | 0

119. Other Pre Specified Outcome: Part A: Titers of Anti-N, Anti-S and Anti-RBD SARS-CoV-2 Antibodies at Baseline
Description: Serum samples were planned to be collected for the determination of anti-drug antibodies using a validated ECL immunoassay. The results for this outcome measure will never be posted.
Time Frame: Baseline (Day 1)
Population: as for outcome 104
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 0 | 0

120. Other Pre Specified Outcome: Part B: Titers of Anti-N, Anti-S and Anti-RBD SARS-CoV-2 Antibodies at Baseline
Description: as for outcome 119
Time Frame: Baseline (Day 1)
Population: as for outcome 104
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 0 | 0

121. Other Pre Specified Outcome: Part C: Titers of Anti-N, Anti-S and Anti-RBD SARS-CoV-2 Antibodies at Baseline
Description: as for outcome 119
Time Frame: Baseline (Day 1)
Population: as for outcome 104
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 0 | 0

122. Other Pre Specified Outcome: Part A: Number of Participants With the Presence of Anti-N SARS-CoV-2 Antibodies at Day 29
Description: Number of participants with the presence of Anti-N SARS-CoV-2 antibodies were planned to be evaluated. The results for this outcome measure will never be posted.
Time Frame: Day 29
Population: as for outcome 104
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 0 | 0

123. Other Pre Specified Outcome: Part B: Number of Participants With the Presence of Anti-N SARS-CoV-2 Antibodies at Day 29
Description: as for outcome 122
Time Frame: Day 29
Population: as for outcome 104
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 0 | 0

124. Other Pre Specified Outcome: Part C: Number of Participants With the Presence of Anti-N SARS-CoV-2 Antibodies at Day 29
Description: as for outcome 122
Time Frame: Day 29
Population: as for outcome 104
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 0 | 0

125. Other Pre Specified Outcome: Part A: Titers of Anti-N SARS-CoV-2 Antibodies at Day 29
Description: as for outcome 119
Time Frame: Day 29
Population: as for outcome 104
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV
Number analyzed (Participants) | 0 | 0

126. Other Pre Specified Outcome: Part B: Titers of Anti-N SARS-CoV-2 Antibodies at Day 29
Description: as for outcome 119
Time Frame: Day 29
Population: as for outcome 104
Arm/Group | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM
Number analyzed (Participants) | 0 | 0

127. Other Pre Specified Outcome: Part C: Titers of Anti-N SARS-CoV-2 Antibodies at Day 29
Description: as for outcome 119
Time Frame: Day 29
Population: as for outcome 104
Arm/Group | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious AEs and SAEs were collected up to Week 24 in Part A; and up to Week 36 in Parts B and C of the study
Description: Safety Population consisted of all randomized participants who were exposed to study intervention.
Arm/Group | Part A-Sotrovimab Gen1: 500 mg IV | Part A- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IV | Part B- Sotrovimab Gen2: 500 mg IM | Part C- Sotrovimab Gen2: 500 mg IV | Part C- Sotrovimab Gen2: 250 mg IM
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/22 | 0/84 | 0/82 | 0/79 | 1/78
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/22 | 1/84 | 2/82 | 2/79 | 3/78
Other Adverse Events (participants affected / at risk) | 0/8 | 6/22 | 8/84 | 20/82 | 16/79 | 16/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A-Sotrovimab Gen1: 500 mg IV (N=8) | Part A- Sotrovimab Gen2: 500 mg IV (N=22) | Part B- Sotrovimab Gen2: 500 mg IV (N=84) | Part B- Sotrovimab Gen2: 500 mg IM (N=82) | Part C- Sotrovimab Gen2: 500 mg IV (N=79) | Part C- Sotrovimab Gen2: 250 mg IM (N=78)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Coronavirus pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A-Sotrovimab Gen1: 500 mg IV (N=8) | Part A- Sotrovimab Gen2: 500 mg IV (N=22) | Part B- Sotrovimab Gen2: 500 mg IV (N=84) | Part B- Sotrovimab Gen2: 500 mg IM (N=82) | Part C- Sotrovimab Gen2: 500 mg IV (N=79) | Part C- Sotrovimab Gen2: 250 mg IM (N=78)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia Oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uvulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — General disorders and administration site conditions
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — General disorders and administration site conditions
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (13) | 0 (0) | 2 (2) — General disorders and administration site conditions
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — General disorders and administration site conditions
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT04779879/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT04779879/SAP_001.pdf